CLINICAL TRIAL: NCT02510014
Title: An Open-Label, Long-Term Safety and Tolerability Study of Depot Buprenorphine (RBP-6000) in Treatment-Seeking Subjects With Opioid Use Disorder
Brief Title: Safety and Tolerability Study of Depot Buprenorphine in Treatment Seeking Subjects With Opioid Use Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RB-US-13-0003
Record Dates: First submitted 2015-07-20; First posted 2015-07-28 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Opioid Use Disorder; Opioid-related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination; Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Roll-over Subjects (Experimental): Subjects who completed RB-US-13-0001 received SUBOXONE sublingual film during the Run-In period, followed by an initial open-label injection of 300 mg RBP-6000. Participants continued with monthly injections of either 300 mg or 100 mg (based on judgement of the Investigator) for a total of 6 months in the Treatment period.
  Interventions: Drug: SUBOXONE sublingual film; Drug: RBP-6000
- De Novo Subjects (Experimental): Subjects who did not participate in RB-US-13-0001 received SUBOXONE sublingual film during the Run-In period, followed by an initial open-label injection of 300 mg RBP-6000. Participants continued with monthly injections of either 300 mg or 100 mg (based on judgement of the Investigator) for a total of 12 months in the Treatment period.
  Interventions: Drug: SUBOXONE sublingual film; Drug: RBP-6000

INTERVENTIONS:
Drug: SUBOXONE sublingual film — SUBOXONE (buprenorphine sublingual film) is used for induction therapy on Days -14 to -12. Participants then complete a 4-to-11 day sublingual film dose adjustment at doses ranging from 8 mg to 24 mg sublingual film prior to starting the Treatment Period.
  Other Names: SUBOXONE; buprenorphine
Drug: RBP-6000 — Injections administered subcutaneously every 28 days on alternate sides of participant's abdomen starting at 300 mg. Subsequent doses of RBP-6000 could be adjusted down to 100 mg with the possibility of adjusting back up to 300 mg based on the medical judgment of the investigator. De novo subjects receive up to 12 injections and roll-over subjects receive up to 6 injections.
  Other Names: Atrigel buprenorphine

SUMMARY:
A multi-center, open-label, long-term safety study in which approximately 600 subjects diagnosed with opioid use disorder will be enrolled. Following a screening period, all subjects will receive run in SUBOXONE sublingual film followed by an initial injection of open-label high dose (300 mg) RBP-6000. The RBP-6000 monthly injection dose can be adjusted to low dose (100 mg), and back to high dose, based on the medical judgment of the Investigator. Subjects will participate in the study for either 6 or 12 months.

DETAILED DESCRIPTION:
Approximately 600 subjects diagnosed with opioid use disorder will be enrolled; approximately 300 subjects who completed the randomized,double-blind, placebo-controlled study NCT02357901 (RB-US-13-0001) ('roll-over' participants), and approximately 300 subjects who did not participate in study RB-US-13-0001 ('de novo' participants). Following informed consent and completion of screening procedures, all subjects will receive SUBOXONE sublingual film, titrated to response.

After 4-14 days of SUBOXONE sublingual film treatment, subjects will be evaluated for enrollment into the study. Eligible subjects will receive 300 mg RBP-6000 as an initial dose, followed by monthly injections of 100 mg or 300 mg RBP-6000, based on the medical judgment of the investigator.

Subjects who participated in study RB-US-13-0001 ('roll-over' participants) will receive monthly injections for up to 6 months. Subjects who did not participate in study RB-US-13-0001 ('de novo' participants) will receive monthly injections for up to12 months.

At all injection visits continuous electrocardiogram recordings and pulse oximetry will be collected prior to injection and at least 4 hours after injection. Subjects will return to the clinic every 1-4 weeks for laboratory tests, complete study questionnaires, adverse event and injection site assessments.

ELIGIBILITY:
Inclusion Criteria:

De novo subjects:

* Seeking treatment for opioid use disorder (OUD) and for the previous 3 months meet the Diagnostic and Statistical Manual 5 (DSM-5) criteria for moderate or severe OUD
* Appropriate candidate for opioid partial-agonist treatment
* BMI between 18 and 35, inclusive

Roll-over subjects:

* Completed RB-US-13-0001

Exclusion Criteria:

De novo subjects:

* Current diagnosis, other than OUD, requiring chronic opioid treatment
* Current substance use disorder with regard to substances other than opioids, cocaine, cannabis, tobacco or alcohol
* Received medication-assisted treatment for OUD in the 90 days prior to informed consent
* Use (within past 30 days prior to informed consent) or positive urine drug screen (UDS) at screening for barbiturates, benzodiazepines,methadone or buprenorphine
* Treatment for OUD required by court order
* History of recent suicidal ideation or attempt

Roll over subjects:

* Experienced major protocol deviations or adverse events in RB-US-13-0001 which could potentially compromise subject safety
* Discontinued early from study RB-US-13-0001

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 775 (Actual)
Dates: Start 2015-07-27 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Director Clinical Development, Study Director — Indivior Inc.
Locations (42):
- United States (42):
  - Haleyville Clinical Research, Haleyville, Alabama
  - Boyett Health Services, Hamilton, Alabama
  - Woodland International Research Group, Little Rock, Arkansas
  - Collaborative Neuroscience Network, Garden Grove, California
  - Behavioral Research Specialists, Glendale, California
  - Synergy Clinical Research Center, National City, California
  - Pacific Research Partners, Oakland, California
  - North County Clinical Research, Oceanside, California
  - Neuropsychiatric Research Center of Orange County, Orange, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Amit Vijapura, Jacksonville, Florida
  - Sarkis Clinical Trials, Lake City, Florida
  - Meridien Research, Lakeland, Florida
  - Innovative Clinical Research, Lauderhill, Florida
  - Florida Clinical Research Center, Maitland, Florida
  - Try Research, Maitland, Florida
  - Scientific Clinical Research, North Miami, Florida
  - Research Centers of America, Oakland Park, Florida
  - Atlanta Institute of Medicine and Research, Alpharetta, Georgia
  - Phoenix Medical Research, Prairie Village, Kansas
  - Louisiana Research Associates, New Orleans, Louisiana
  - Louisiana Clinical Research, Shreveport, Louisiana
  - Stanley Street Treatment and Resources, Fall River, Massachusetts
  - Adams Clinical Trials, Watertown, Massachusetts
  - Precise Research Centers, Inc., Flowood, Mississippi
  - St Louis Clinical Trials, St Louis, Missouri
  - Altea Research, Las Vegas, Nevada
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - The Medical Research Network, LLC, New York, New York
  - Neuro-behavioral Clinical Research, Canton, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Charak Clinical Research Center, Garfield Heights, Ohio
  - Oklahoma Clinical Research Center, Oklahoma City, Oklahoma
  - Pahl Pharmaceutical Professionals, Oklahoma City, Oklahoma
  - CODA, Portland, Oregon
  - Tipton Medical and Diagnostic Center aka Clinical Research Associates of Central PA, Altoona, Pennsylvania
  - UPenn Treatment Research Center, Philadelphia, Pennsylvania
  - Carolina Clinical Trials, Charleston, South Carolina
  - Pillar Clinical Research, Dallas, Texas
  - InSite Clinical Research, DeSoto, Texas
  - Aspen Clinical Research, LLC, Orem, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rutrick D, Learned SM, Boyett B, Hassman D, Shinde S, Zhao Y. 18-Month efficacy and safety analysis of monthly subcutaneous buprenorphine injection for opioid use disorder: Integrated analysis of phase 3 studies. J Subst Use Addict Treat. 2023 Nov;154:209155. doi: 10.1016/j.josat.2023.209155. Epub 2023 Aug 30. PMID 37657559
- [Derived] Craft WH, Tegge AN, Keith DR, Shin H, Williams J, Athamneh LN, Stein JS, Chilcoat HD, Le Moigne A, DeVeaugh-Geiss A, Bickel WK. Recovery from opioid use disorder: A 4-year post-clinical trial outcomes study. Drug Alcohol Depend. 2022 May 1;234:109389. doi: 10.1016/j.drugalcdep.2022.109389. Epub 2022 Mar 9. PMID 35287034

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 994 subjects were screened by 39 sites, and of those, 775 subjects entered the run-in period receiving at least 1 dose of SUBOXONE (508 de novo subjects and 267 roll-over subjects).
Period: Run-In Period (Days -14 to Day -1)
Arm/Group | De Novo Subjects | Roll-over Subjects
Started (Received at least one dose of SUBOXONE sublingual film.) | 508 | 267
Completed | 412 | 257
Not Completed | 96 | 10
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal symptoms | 1 | 0
Not completed — Lost to Follow-up | 44 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 22 | 3
Not completed — Withdrawn by the investigator | 7 | 1
Not completed — Protocol Violation | 2 | 0
Not completed — Other | 19 | 1
Period: Treatment Period
Arm/Group | De Novo Subjects | Roll-over Subjects
Started | 412 | 257
Completed | 206 | 200
Not Completed | 206 | 57
Not completed — Adverse Event | 11 | 4
Not completed — Withdrawal symptoms | 3 | 0
Not completed — Lost to Follow-up | 80 | 19
Not completed — Physician Decision | 5 | 0
Not completed — Withdrawal by Subject | 67 | 24
Not completed — Withdrawn by the investigator | 7 | 1
Not completed — Protocol Violation | 4 | 4
Not completed — Incarceration, pregnancy, misc | 29 | 5

BASELINE CHARACTERISTICS:
Population: Safety analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | De Novo Subjects | Roll-over Subjects | Total
Number analyzed (Participants) | 412 | 257 | 669
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (12.10) | 41.6 (11.07) | 39.6 (11.81)
Age, Customized [Count of Participants; unit: Participants]
  >=18 to <30 years | 122 | 40 | 162
  >=30 to <45 years | 157 | 114 | 271
  >=45 to <60 years | 107 | 89 | 196
  >= 60 to < 65 years | 25 | 14 | 39
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 88 | 237
  Male | 263 | 169 | 432
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 16 | 59
  Not Hispanic or Latino | 369 | 241 | 610
Race [Count of Participants; unit: Participants]
  White | 295 | 167 | 462
  Black or African American | 107 | 85 | 192
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 2 | 0 | 2
  Multiple | 2 | 2 | 4
  Other | 4 | 0 | 4
Weight [Mean (Standard Deviation); unit: kg] | 75.49 (14.658) | 78.43 (18.097) | 76.62 (16.117)
Waist-to-Hip Ratio [Mean (Standard Deviation); unit: ratio] — Waist-to-hip ratio is the ratio of the waist circumference to hip circumference (calculated by dividing the waist circumference by the hip circumference). It is a measurement of abdominal fat distribution. Population: Records for one participant were missing baseline waist-to-hip ratio.
  ratio
    number analyzed (Participants) | 411 | 257 | 668
    (all) | 0.91 (0.086) | 0.90 (0.083) | 0.90 (0.085)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.38 (4.286) | 26.14 (5.067) | 25.67 (4.613)
Tobacco use [Count of Participants; unit: Participants]
  Never | 40 | 23 | 63
  Former | 18 | 12 | 30
  Current | 354 | 222 | 576
Caffeine use [Count of Participants; unit: Participants]
  Never | 33 | 21 | 54
  Former | 13 | 7 | 20
  Current | 365 | 229 | 594
  Missing data | 1 | 0 | 1
Alcohol use [Count of Participants; unit: Participants]
  Never | 122 | 48 | 170
  Former | 97 | 65 | 162
  Current | 193 | 144 | 337

OUTCOME MEASURES:

1. Primary Outcome: Participants With Treatment-Emergent Adverse Events (TEAE) During the Treatment Period
Description: TEAE=any untoward medical occurrence that develops or worsens in severity after dispensation of the study drug and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= a marked limitation in activity. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Day 1 to Week 49 (De novo arm); Day 1 to Week 25 (Roll-over arm)
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | De Novo Subjects | Roll-over Subjects
Number analyzed (Participants) | 412 | 257
Participants
  >=1 TEAE | 302 | 145
  >=1 TEAE related to study drug | 172 | 61
  >=1 serious TEAE | 16 | 9
  >=1 serious study treatment-related TEAE | 0 | 0
  Death | 0 | 0
  >=1 severe TEAE | 36 | 7
  TEAE leading to study treatment discontinuation | 13 | 4
  TEAE leading to dose reduction | 29 | 17

2. Primary Outcome: Percentage Change From Baseline to End of Study (Weeks 25 and 49) in Vital Signs
Description: Vital signs include
  * systolic blood pressure (mmHg)
  * diastolic blood pressure (mmHg)
  * respiratory rate (breaths/minute)
  * weight (kg)
  * body mass index (kg/m^2)
  * waist-to-hip ratio
  Baseline is defined as the last non-missing value prior to subcutaneous injection of RBP-6000 on Day 1.
Time Frame: Baseline (Day 1 predose) End of Study: Week 49 (De novo arm); Week 25 (Roll-over arm)
Population: Safety analysis set of participants with both a baseline and end of study reading
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | De Novo Subjects | Roll-over Subjects
Number analyzed (Participants) | 206 | 198
percentage change from baseline
  Systolic blood pressure | 0.2 (11.69) | 1.3 (11.25)
  Diastolic blood pressure | 0.1 (13.97) | 1.6 (12.49)
  Respiratory rate: number analyzed (Participants) | 205 | 198
  Respiratory rate | -1.2 (11.11) | 1.0 (11.02)
  Body weight: number analyzed (Participants) | 206 | 197
  Body weight | 1.52 (10.651) | -0.94 (6.497)
  Body mass index: number analyzed (Participants) | 206 | 197
  Body mass index | 1.53 (10.657) | -0.93 (6.507)
  Waist-to-hip ratio: number analyzed (Participants) | 204 | 195
  Waist-to-hip ratio | 1.828 (11.1698) | 1.015 (8.1150)

3. Primary Outcome: Shifts in Suicidality Using the Columbia Suicide Severity Rating Scale (C-SSRS) From Baseline to Most Severe Assessment During the Treatment Period
Description: The C-SSRS asks questions of study participants regarding whether they had suicidal ideation and/or suicidal behavior since the last visit using the electronic version of the scale. Only the most severe assessment is reported in this summary. Participants who experienced suicidal ideation and suicidal behavior are only summarized in the suicidal behavior since behavior is more severe than ideation.
  C-SSRS baseline version was completed during the screening visit. C-SSRS 'since-last-visit' version was completed weekly for the first month and at least every month until the end of the study.
  Shift table category titles are structured as: baseline category/treatment category. The category 'No Suicidal Ideation or Behaviour' has been abbreviated as 'No Suicidal I or B'.
Time Frame: Baseline (Screening visit, days -21 to -15), End of Study: Week 49 (De novo arm); Week 25 (Roll-over arm)
Population: Safety population. Four de novo subjects and one roll-over subject are not reported because they used the C-SSRS baseline version throughout the study.
Measure: Count of Participants; unit: Participants
Arm/Group | De Novo Subjects | Roll-over Subjects
Number analyzed (Participants) | 408 | 256
Participants
  No Suicidal I or B / No Suicidal I or B | 307 | 252
  No Suicidal I or B / Suicidal Ideation | 10 | 1
  No Suicidal I or B / Suicidal Behaviour | 3 | 1
  Suicidal Ideation / No Suicidal I or B | 46 | 1
  Suicidal Ideation / Suicidal Ideation | 7 | 1
  Suicidal Ideation / Suicidal Behaviour | 3 | 0
  Suicidal Behaviour / No Suicidal I or B | 28 | 0
  Suicidal Behaviour / Suicidal Ideation | 2 | 0
  Suicidal Behaviour / Suicidal Behaviour | 2 | 0

4. Primary Outcome: Worst Local Injection Site Pain From Injections as Measured by Participant-Reported Visual Analog Scale (VAS)
Description: Injection site pain as measured by participant-reported VAS. The participant-reported VAS for injection site pain was measured on a 100 mm scale with 'no pain' at 0 mm and 'strongest pain ever' at 100 mm (total scale of 0-100). Participants marked where along the scale reflected their localized injection pain.
  The injection site pain VAS scores were obtained (after the completion of the injection) within 1 minute and at 5, 10, 15, 30 and 60 minutes (+- 5 minutes). The timing of the injection site pain VAS should have been measured from the end of the injection.
  Data represents the worst pain recorded for each participant across all injections and all VAS records. The mean value is presented.
  De Novo subjects were given injections on Days 1, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281 and 309.
  Roll-over subjects were given injections on Days 1, 29, 57, 85, 113, 141.
Time Frame: De Novo Subjects: Days 1, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281 and 309 Roll-over Subjects: Days 1, 29, 57, 85, 113, 141
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | De Novo Subjects | Roll-over Subjects
Number analyzed (Participants) | 412 | 257
units on a scale
  Injection 1 | 44.0 (29.86) | 33.5 (31.50)
  Injection 2: number analyzed (Participants) | 365 | 249
  Injection 2 | 39.8 (31.98) | 32.7 (31.59)
  Injection 3: number analyzed (Participants) | 342 | 235
  Injection 3 | 38.9 (32.14) | 30.2 (32.09)
  Injection 4: number analyzed (Participants) | 314 | 221
  Injection 4 | 33.6 (32.86) | 31.3 (31.72)
  Injection 5: number analyzed (Participants) | 295 | 210
  Injection 5 | 30.6 (30.96) | 32.2 (31.25)
  Injection 6: number analyzed (Participants) | 280 | 202
  Injection 6 | 30.5 (31.89) | 30.5 (30.88)
  Injection 7: number analyzed (Participants) | 264 | 0
  Injection 7 | 28.9 (32.13) |
  Injection 8: number analyzed (Participants) | 251 | 0
  Injection 8 | 28.6 (30.21) |
  Injection 9: number analyzed (Participants) | 242 | 0
  Injection 9 | 30.2 (33.96) |
  Injection 10: number analyzed (Participants) | 232 | 0
  Injection 10 | 31.8 (33.16) |
  Injection 11: number analyzed (Participants) | 228 | 0
  Injection 11 | 25.8 (30.71) |
  Injection 12: number analyzed (Participants) | 219 | 0
  Injection 12 | 24.7 (28.22) |

5. Secondary Outcome: Change From Baseline in the Clinical Opiate Withdrawal Scale (COWS) at End of Study (Weeks 25 and 49)
Description: COWS is an 11-item instrument used to assess signs and symptoms of opioid withdrawal. The score is the sum of the responses for a total range of 0-48. The COWS is commonly used by clinicians treating patients with buprenorphine to monitor the severity of withdrawal. COWS scores below 5 are considered not indicative of withdrawal. Scores from 5 to 12 are considered mild withdrawal; from 13 to 24 moderate withdrawal; 25 to 36 moderately severe withdrawal, and 37-48 severe withdrawal. Negative change from baseline values indicate a lessening of withdrawal symptoms.
  Baseline was defined as the last non-missing value prior to subcutaneous injection on Day 1. Baseline value is reported as an observed actual value. Weeks 25 and 49 represent change from baseline values.
Time Frame: Baseline (Day 1 predose), End of Study: Week 49 (De novo arm); Week 25 (Roll-over arm)
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | De Novo Subjects | Roll-over Subjects
Number analyzed (Participants) | 412 | 257
units on a scale
  Baseline (actual value) | 2.1 (2.43) | 1.5 (1.98)
  Change from baseline: Week 25: number analyzed (Participants) | 267 | 199
  Change from baseline: Week 25 | -1.0 (2.61) | -0.3 (2.37)
  Change from baseline: Week 49: number analyzed (Participants) | 202 | 0
  Change from baseline: Week 49 | -1.0 (2.41) |

6. Secondary Outcome: Change From Baseline in the Subjective Opiate Withdrawal Scale (SOWS) at End of Study (Weeks 25 and 49)
Description: The Subjective Opiate Withdrawal Scale (SOWS) contains 16 symptoms whose intensity the participant rates on a scale of 0 (not at all) to 4 (extremely) for a full scale of 0 (no withdrawal symptoms) to 64 (extreme withdrawal symptoms). Negative change from baseline values indicate a lessening of withdrawal symptoms.
  Baseline was defined as the last non-missing value prior to subcutaneous injection on Day 1. Baseline value is reported as an observed actual value. Weeks 25 and 49 represent change from baseline values.
Time Frame: Baseline (Day 1 predose), End of Study: Week 49 (De novo arm); Week 25 (Roll-over arm)
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | De Novo Subjects | Roll-over Subjects
Number analyzed (Participants) | 412 | 257
units on a scale
  Baseline (actual value) | 3.8 (5.27) | 2.8 (5.44)
  Change from baseline: Week 25: number analyzed (Participants) | 271 | 200
  Change from baseline: Week 25 | -1.1 (6.63) | 1.1 (7.17)
  Change from baseline: Week 49: number analyzed (Participants) | 203 | 0
  Change from baseline: Week 49 | -1.6 (5.05) |

7. Secondary Outcome: Change From Baseline in the Opioid Craving Visual Analog Scale (VAS) at End of Study (Weeks 25 and 49)
Description: The opioid craving scale was a 100 mm scale with 'no craving' indicated by 0 mm and 'strongest craving ever' indicated by 100 mm. Participants marked where along the scale reflected their craving for opioids.
  Baseline was defined as the last non-missing value prior to subcutaneous injection on Day 1. Baseline value is reported as an observed actual value. Weeks 25 and 49 represent change from baseline values.
Time Frame: Baseline (Day 1 predose), End of Study: Week 49 (De novo arm); Week 25 (Roll-over arm)
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | De Novo Subjects | Roll-over Subjects
Number analyzed (Participants) | 412 | 257
units on a scale
  Baseline (actual value) | 5.9 (10.59) | 4.4 (9.62)
  Change from baseline: Week 25: number analyzed (Participants) | 271 | 200
  Change from baseline: Week 25 | -0.2 (16.19) | 4.2 (16.77)
  Change from baseline: Week 49: number analyzed (Participants) | 203 | 0
  Change from baseline: Week 49 | -2.0 (10.83) |

8. Secondary Outcome: Cumulative Distribution Function (CDF) of the Percentage Abstinence Collected From Week 1 Through End of Study (Weeks 25 and 49)
Description: Participants' self-reported illicit opioid drug use from the timeline followback (TLFB) interview and results from the urine drug screens (UDS) for opioids were combined into a single endpoint. Opioids assessed included codeine, hydrocodone, hydromorphone, methadone, morphine, opiates, oxycodone, and oxymorphone (by UDS) and amphetamine/methadone, buprenorphine, methadone, and opioids in the TLFB.
  Data represent the count of participants at various percentage abstinence levels. Abstinence was defined as urine samples being negative for opioids AND negative self-reports (obtained from Timeline Followback (TLFB) interviews) for illicit opioid use. The endpoint was based on visits in which paired urine samples and self-reports were expected for each subject as specified in the schedule of events. All missing reports for opioids were considered nonnegative.
Time Frame: Weekly during Month 1, Every other week from Month 2-6, Monthly from Month 7-12. De novo arm stopped at Week 49. Roll-over arm stopped at Week 25
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | De Novo Subjects | Roll-over Subjects
Number analyzed (Participants) | 412 | 257
Participants
  >=0% | 412 | 257
  >=10% | 315 | 206
  >=20% | 278 | 200
  >=30% | 239 | 189
  >=40% | 217 | 159
  >=50% | 187 | 150
  >=60% | 166 | 137
  >=70% | 132 | 110
  >=80% | 98 | 96
  >=90% | 62 | 74
  =100% | 32 | 47

ADVERSE EVENTS:
Time Frame: Day 1 to Week 49 for De Novo arm Day 1 to Week 25 for the Roll-over arm
Arm/Group | De Novo Subjects | Roll-over Subjects
All-Cause Mortality (participants affected / at risk) | 0/412 | 0/257
Serious Adverse Events (participants affected / at risk) | 16/412 | 9/257
Other Adverse Events (participants affected / at risk) | 146/412 | 42/257
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | De Novo Subjects (N=412) | Roll-over Subjects (N=257)
Cellulitis (Infections and infestations) | 2 | 1
Abscess limb (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Escherichia pyelonephritis (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0
Prostatic abscess (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Adjustment disorder with mixed anxiety and depressed mood (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Mania (Psychiatric disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Gallbladder perforation (Hepatobiliary disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | De Novo Subjects (N=412) | Roll-over Subjects (N=257)
Constipation (Gastrointestinal disorders) | 47 | 9
Nausea (Gastrointestinal disorders) | 37 | 10
Injection site pain (General disorders) | 39 | 7
Insomnia (Psychiatric disorders) | 27 | 10
Headache (Nervous system disorders) | 31 | 5
Nasopharyngitis (Infections and infestations) | 24 | 6
Injection site erythema (General disorders) | 22 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Proposed publications shall be submitted to Sponsor 30 days prior to submission for publication, and may be withheld for an additional period, up to 90 days, to allow Sponsor to file patent applications. If a multi-center publication isn't submitted for publication within 12 months of the conclusion of the Study at all sites, or is published in a shorter period, the results from the institution's site may be published individually.

DOCUMENTS (6):
  • Study Protocol: Original (2015-04-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT02510014/Prot_000.pdf
  • Study Protocol: Amendment 1 (2015-08-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT02510014/Prot_001.pdf
  • Study Protocol: Amendment 2 (2015-09-11): https://cdn.clinicaltrials.gov/large-docs/14/NCT02510014/Prot_002.pdf
  • Study Protocol: Amendment 3 (2016-03-25): https://cdn.clinicaltrials.gov/large-docs/14/NCT02510014/Prot_003.pdf
  • Statistical Analysis Plan (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT02510014/SAP_004.pdf
  • Study Protocol: Amendment 4 (2016-08-04): https://cdn.clinicaltrials.gov/large-docs/14/NCT02510014/Prot_005.pdf